CLINICAL TRIAL: NCT05123053
Title: Amifampridine for the Treatment of Transient Vocal Weakness After OnabotulinumtoxinA Injection for Spasmodic Dysphonia
Brief Title: Firdapse for Post-BOTOX Vocal Weakness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD-DAP-01
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-02

CONDITIONS: Vocal Weakness(Post-BOTOX Injection)
Keywords: BOTOX; Onabotulinumtoxin; Spasmodic Dysphonia
MeSH Terms: conditions — Dysphonia | interventions — Amifampridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): subjects will be given active drug and titrated up in 10mg increments (with max single dose being 30mg) until a change or drug side effect is noticed.
  Interventions: Drug: Amifampridine

INTERVENTIONS:
Drug: Amifampridine — 10mg tablet
  Other Names: Firdapse

SUMMARY:
Botox injections into the thyroarytenoid muscle are a predictable and effective treatment for SD, but typically result in transient symptoms of voice weakness and breathiness during the first 2-3 weeks after injection. Investigators hypothesize that voice weakness and breathiness after Botox treatment can be alleviated using amifampridine.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD) is a dystonia which results in vocal breaks. The mainstay of treatment involves injections using Botox (onabotulinumtoxinA), a neuromuscular blocker which inhibits pre-synaptic release of acetylcholine into the neuromuscular junction. Botox injections into the thyroarytenoid muscle are a predictable and effective treatment for SD, but typically result in transient symptoms of voice weakness and breathiness during the first 2-3 weeks after injection. These symptoms can be present for even longer if Botox is over- dosed.

Investigators hypothesize that these initial, transient symptoms of voice weakness and breathiness after Botox treatment can be alleviated using amifampridine which acts at the neuromuscular junction to increase synaptic presence of the neurotransmitter acetylcholine. In these initial studies, investigators will look at patients who have significant breathiness following an injection.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age.
2. Capable of providing informed consent.
3. Confirmed physician diagnosis of spasmodic dysphonia.
4. Receives onabotulinumtoxinA for treatment of their spasmodic dysphonia.
5. Experiences significant breathiness ± 5 days following their injection.
6. If sexually active and of childbearing potential, willing to use an acceptable method of contraception (as noted below) from screening visit until 3 months after the last dose of investigational product.

A.NOTE: No adequate clinical data on exposed pregnancies are available for amifampridine. No nonclinical safety data are available regarding the effects of amifampridine on reproductive function. Amifampridine phosphate should not be used during pregnancy. It is unknown whether amifampridine is excreted in human breast milk. The excretion of amifampridine in milk has not been studied in animals. Amifampridine phosphate should not be used during breastfeeding. Acceptable methods of birth control include:

1. Hormonal contraception (e.g., oral contraceptive, transdermal contraceptive, contraceptive implant, or injectable hormonal contraceptive) for at least 3 months prior to study drug administration, throughout the study, and for 3 months after the last dose of study drug.
2. Double-barrier birth control (e.g., a combination of male condom with either cap, diaphragm, or sponge together with spermicide) starting at the Screening visit, throughout the study, and for at least 4 weeks after the last dose of study drug. NOTE: Use of a male and female condom simultaneously is NOT an acceptable method of double-barrier birth control.
3. Intrauterine contraception/device starting at the Screening visit, throughout the study, and for 3 months after the last dose of study drug.
4. Total abstinence from sexual intercourse (only acceptable if it is the preferred and usual lifestyle of the subject) for at least 1 complete menstrual cycle prior to the Screening visit, throughout the study, and for 3 months after the last dose of study drug.
5. Maintenance of a monogamous relationship with a male partner who has been surgically sterilized by vasectomy.

B. NOTE: Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception.

Exclusion Criteria:

1. History of epilepsy and/or on medication/treatment for seizures (such as but not limited to valproic acid, lamotrigine, topiramate, carbamazepine, and phenytoin); or, on certain medications that may lower seizure threshold, such as:

   1. anaesthetic drugs (propofol),
   2. antibiotics (penicillins, cephalosporins, imipenem),
   3. some antidepressants (clomipramine, bupropion, and maprotiline),
   4. antipsychotics (clozapine, chlorpromazine),
   5. bronchodilators (aminophylline, theophylline),
   6. Immunomodifiers (cyclosporine), and
   7. Narcotic analgesics (pethidine, fentanyl).
2. Any SGOT, SGPT that are more than 3x upper limit of normal; and, creatinine that is greater than 2.1
3. Women who are pregnant, expecting to get pregnant, or breastfeeding.
4. Any condition that, in the view of the Principal Investigator, places the subject at risk, or subjects with poor treatment compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Voice Handicap Index-10 | over 2 months
  VHI-10 is a scale used to assess the severity of problematic symptoms associated with the voice. It is a series of 10 questions. Each questions is answered using numbers 0-4, with 0 meaning the patient never has a problem with that symptom; and, 4 meaning the patient always has a problem with that symptom.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Rivner, MD, Principal Investigator — Charbonnier Professor Emeritus of Neurology
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No